CLINICAL TRIAL: NCT00722306
Title: A Phase One Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism And Excretion Of [14C] PD 0200390 In Six Healthy Male Volunteers
Brief Title: A Study To Investigate The Absorption, Metabolism And Excretion Of [14C] PD 0200390 In Six Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4251072
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Insomnia
Keywords: non-restorative; sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — (1-aminomethyl-3,4-dimethylcyclopentyl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A425 (Experimental): A425 Treated
  Interventions: Drug: PD 0200390

INTERVENTIONS:
Drug: PD 0200390 — Extemporaneous solution of C14 Labelled PD 0200390 60 mg single dose

SUMMARY:
To determine the mass balance of PD 0200390

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* unhealthy, or concomitant meds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Radioactivity parameters in plasma and whole blood - Cmax , Tmax , AUCinf, AUClast, t1/2, CL/F and V/F and Total 14C data in blood, urine and feces | 2 days

SECONDARY OUTCOMES:
% urinary recovery | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4251072&StudyName=A425%20Mass%20Balance%20Study